CLINICAL TRIAL: NCT05212376
Title: The Impact of Foot Massage Applied to Menopausal Women on Anxiety, Fatigue and Sleep Level
Brief Title: Foot Massage for Women With Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Çiğdem KARAKAYALI AY, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/2497
Record Dates: First submitted 2022-01-11; First posted 2022-01-28 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Menopausal Women
Keywords: Menopause; Fatigue; Anxiety; Sleep; Foot massage
MeSH Terms: conditions — Fatigue; Anxiety Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot massage (Experimental): Foot massage (reflexology) is an application that allows the individual to relax, reduce stress, and thus restore the balance of the body by stimulating the nerve cells in the legs.It is stated that reflexology is an effective complementary treatment method that can help the body relax, reduce the symptoms of menopause by affecting the nervous and endocrine system, and thus create a smooth transition to the menopausal period.
  Interventions: Other: Foot massage
- Control group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: Foot massage — Foot massage is applied in the form of pressure, rubbing and stimulation with special hand and finger techniques to reflex - warning points corresponding to all regions, organs and systems in the body. It is applied by applying pressure to all reflex points in the area from the toes to the ankles.
  In the study, a quiet and comfortable environment will be prepared at a room temperature of approximately 23-26 0C, and techniques that reveal the relaxing and calming effect of the massage will be selected. Thumb compression, slapping, patting, rubbing and squeezing movements are planned to be applied for a total of 20 minutes, 10 minutes on each foot, at the same time every day for 7 days.
  Other Names: Reflexology
  Arms: Foot massage

SUMMARY:
This study will be carried out to determine the effect of foot massage applied to menopausal women on anxiety, fatigue and sleep levels. This randomized controlled study will be conducted with 70 women (35 experimental, 35 control) residing in a village in northern Turkey. In the study, women in the experimental group will be given foot massage once a day for 7 days. No intervention will be applied to the women in the control group. Research data will be collected using "Personal Information Form", "Fatigue Severity Scale" and "Beck Anxiety Inventory". Descriptive statistics (number, percentage distribution, median and Q1-Q3), chi-square test, Mann Whitney-U test and Wilcoxon test will be used in the analysis of the data.

DETAILED DESCRIPTION:
The population of the study was planned to be composed of menopausal women residing in a village in the north of Turkey. Menopausal women residing in the village were reached from the records of the health unit of the participants. The number of people to be included in the sample of the study was determined by power analysis. G*power 3.1.9.2 program was used in the study. According to the calculations made, the minimum sample size of the study was 0.40, the error level was 0.05, and the population representativeness was 0.95 to 64 women (32 experiment, 32 control). Considering the possible data losses (10%), 70 women (35 experimental, 35 control) were planned to be included in the study. It was planned to include women who are literate, open to communication, and have naturally entered menopause in the last 1 year. The data are planned to be collected by the researchers through face-to-face interviews at the homes of menopausal women residing in a village in northern Turkey between 01-30 November 2021.

Experimental group Menopausal women in the experimental group will be met at the first interview at their home, the participants will be informed about the method and their written consent will be obtained. Pre-test data will be obtained by filling in the personal information form, "Fatigue Severity Scale" and "Beck Anxiety Inventory" before the foot massage. The same researcher will plan to give women a foot massage once a day for 7 days. It is anticipated that the foot massage application will take a total of 20 minutes on both feet. On the last day (7th day), 30 minutes after the foot massage, FSS and BAI will be applied again and the final test data will be obtained.

Control group Menopausal women in the control group will be met at the first interview at their homes, the participants will be informed about the method and their written consent will be obtained. It will be planned to obtain the pre-test data by filling in the "Fatigue Severity Scale" and "Beck Anxiety Inventory". No intervention will be applied to the women in the control group. A second home visit will be made one week after the pre-test data are received and the post-test data will be obtained.

The initiative will be implemented by an internationally certified research midwife academic (N.G.) after a training on foot massage (16 hours). It is planned to create a quiet and comfortable environment at a room temperature of approximately 23-26 C, and to choose techniques that reveal the relaxing and calming effect of the massage. Thumb pressure application, slapping, patting, rubbing and squeezing movements will be applied for a total of 20 minutes, 10 minutes on each foot, at the same time every day for 7 days.

To evaluate the fatigue and anxiety levels, pretest and posttest data will be obtained by applying FSS and BAI just before the first foot massage (day 1) and 30 minutes after the last foot massage (day 7).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 53-60 years who have gone through natural or surgical menopause
* Women who can read and write.
* Turkish-speaking women.

Exclusion Criteria:

* Do not be diagnosed with any mental illness.
* Existence of a situation that prevents foot massage application

Ages: 53 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Sleep level in women with menopause | Thumb pressure application, swiping, patting, rubbing and squeezing movements were applied to each foot for a total of 20 minutes for 10 minutes, once at the same time every day for 7 days.
  In order to determine the socio-demographic (age, education, employment, income, family type, etc.), obstetric (pregnancy, abortion, number of children, etc.), health status (chronic illness, drug use, etc.) and sleep patterns of women, the researchers It is a form consisting of 25 questions developed by.

SECONDARY OUTCOMES:
Fatigue level in women with menopause | Thumb pressure application, swiping, patting, rubbing and squeezing movements were applied to each foot for a total of 20 minutes for 10 minutes, once at the same time every day for 7 days.
  The scales consist of 9 items. Each item is scored as "1=Strongly disagree, 2= Disagree, 3=Tend not to agree, 4=Hesitant, 5=Tend to disagree, 6=Agree, 7=Definitely agree". The person is asked to select the option that suits them best. The total score is found by the average of 9 questions. A high score indicates an increased degree of fatigue.
Anxiety level in women with menopause | Thumb pressure application, swiping, patting, rubbing and squeezing movements were applied to each foot for a total of 20 minutes for 10 minutes, once at the same time every day for 7 days.
  BAI consists of a total of 21 items. The inventory is 4-point Likert type and each item is scored as "0 =None, 1 =Mild, 2 =Moderate, 3 =Severe". A minimum of 0 and a maximum of 63 points can be obtained from the inventory. An increase in the scores obtained from the inventory indicates that the level of anxiety also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay GÖKBULUT, Principal Investigator — Department of Midwifery, Faculty of Health Sciences, Çankırı Karatekin University; Emine İBİCİ AKÇA, Principal Investigator — Department of Midwifery, Faculty of Health Sciences, Amasya University,; Çiğdem KARAKAYALI AY, Principal Investigator — Department of Midwifery, Faculty of Health Sciences, Inonu University
Locations (1):
- Department of Midwifery, Faculty of Health Sciences Inonu University, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers. Because the institution where the research was conducted does not allow this.

REFERENCES:
- [Background] Gozuyesil E, Baser M. The effect of foot reflexology applied to women aged between 40 and 60 on vasomotor complaints and quality of life. Complement Ther Clin Pract. 2016 Aug;24:78-85. doi: 10.1016/j.ctcp.2016.05.011. Epub 2016 May 24. PMID 27502805
- See also: The effect of foot reflexology applied to women aged between 40 and 60 on vasomotor complaints and quality of life — https://pubmed.ncbi.nlm.nih.gov/27502805/